CLINICAL TRIAL: NCT06981234
Title: Acetazolamide and Tubuloglomerular Feedback in Persons With Type 1 Diabetes: A Randomized Crossover Trial
Brief Title: Acetazolamide in Persons With Type 1 Diabetes - Crossover Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Breakthrough T1D (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 802153-2
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-Controlled, Crossover Trial
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group A (Experimental): 250mg Acetazolamide administered twice a day for 10 weeks followed by Placebo Comparator administered twice a day for 10 weeks.
  Interventions: Drug: Acetazolamide; Drug: Placebo
- Treatment Group B (Experimental): Placebo Comparator administered twice a day for 10 weeks followed by 250mg Acetazolamide administered twice a day for 10 weeks.
  Interventions: Drug: Acetazolamide; Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide is a potent carbonic anhydrase inhibitor that acts on the renal proximal tubule. Through this mechanism, it inhibits proximal tubule sodium reabsorption.
Drug: Placebo — Standard pharmaceutical filler will be capsulated and packaged identically to the acetazolamide.

SUMMARY:
The goal of this study is to learn about the effect of the study drug acetazolamide in individuals with Type 1 Diabetes. Specifically, whether acetazolamide provides benefits to the kidneys while minimizing any side effects of the drug. These changes will be measured by laboratory tests that tell us how well the kidneys are functioning.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Placebo-Controlled, Crossover Trial (RCT) to explore the effects of 250mg acetazolamide in individuals with type 1 diabetes. Participants will be randomized to Treatment Group A or Treatment Group B. Randomization will be blinded, but one of these treatment groups will receive 250mg (milligram) BID (twice daily) of acetazolamide for 10 weeks - receive no study drug for 2 weeks - then receive placebo for 10 weeks; the other will receive placebo for 10 weeks - receive no study drug for 2 weeks - then receive 250mg BID of acetazolamide for 10 weeks. Both participants and study staff will be blinded to the study treatment group with only the research pharmacy staff being unblinded.

To measure mGFR (measured glomerular filtration rate), an Iohexol GFR (glomerular filtration rate) procedure will be completed at the beginning and end of each treatment period. A standard protocol for the procedure will be followed that has been used in multiple studies. Iohexol (Omnipaque 300®) will be used in order to obtain a precise measure of mGRF throughout the course of the test. Iohexol will be prepared by the UCSD (University of California, San Diego) Investigational Drug Services at the ACTRI (Altman Clinical and Translation Research Institute) by drawing up 5mL into a syringe per standard pharmacy protocol. The iohexol will be dispensed to a nurse or research coordinator who will weigh the syringe prior to infusion and again after infusion to assess exact dosage delivered.

A study nurse will insert 1 IV (intravenous) line in the hand or arm for the infusion of iohexol. They will then insert a second IV in the opposite arm for blood collection. Serial blood draws will occur throughout the procedure relative to the time of iohexol infusion. A study nurse will infuse iohexol over a 1-2 minute period, flush with 10mL (milliliter) of normal saline and remove the IV. Blood samples will be collected at the following time points for mGFR analysis:

* -5 minutes (prior to iohexol infusion)
* 2 hours (120 minutes post infusion)
* 4 hours (120 minutes post infusion)
* 6 hours (120 minutes post infusion)

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ≥ 18 years at the time of consent.
2. Individuals able to become pregnant of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Individuals of child bearing potential must agree to use two methods of contraception during the entire study.
3. Individuals able to cause a pregnancy must be willing to use clinically acceptable method of contraception during the entire study.
4. Have a clinical diagnosis of Type 1 Diabetes on a stable medication regimen for at least 3 months.
5. eGFR (estimated glomerular filtration rate) ≥ 45ml/min/1.73m2
6. Serum bicarbonate ≥ 24 meq/L
7. Negative urine toxicology screen.
8. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History of allergic reaction to acetazolamide, another carbonic anhydrase inhibitor, or any of the inactive ingredients in the acetazolamide tablets.
2. Liver disease (clinical diagnosis of cirrhosis by imaging of physician; > 14 drinks/week; AST (Aspartate Transferase), ALT (Alanine Aminotransferase), or total bilirubin > 2 times the upper limit of normal).
3. Serum hemoglobin A1c > 10.0%
4. Serum hemoglobin concentration of <8 g/dL.
5. Use of > 4 anti-hypertensives, or systolic blood pressure >160mm Hg at the screening visit.
6. Use of loop, thiazide or potassium sparing diuretics.
7. A medical condition requiring active surgical or medical intervention whose urgency would preclude participation in this study at the discretion of the site investigator (active cardiac or pulmonary conditions, ongoing ischemia or cardiac symptoms, uncorrected Coronary Artery Disease (CAD) or decompensated congestive heart failure (CHF)).
8. Institutionalized individual (prisoners, patients with signification mental illness, or nursing home residents).
9. Active pregnancy, breastfeeding, or planning to become pregnant during the study period.
10. Current participation in another clinical trial (observational studies are exempted) trial.
11. In the opinion of the investigators, inability to adhere to the study medical regimen or comply with recommendations.
12. Inability or unwillingness to travel to study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in mGFR percent | 10 weeks
  The difference in mGFR percent between acetazolamide versus placebo as measured by the iohexol procedure.
Preservation of Serum Bicarbonate | 10 weeks
  The preservation of serum bicarbonate concentrations at ≥ 20 meq/L (milliequivalents per liter) from pre-dosing to post-treatment iohexol procedure.
Preservation of Serum Potassium | 10 weeks
  The preservation of serum potassium concentrations at ≥ 3.2 meq/L from pre-dosing to post-treatment.
Change is albuminuria | 10 weeks
  The difference in change in albuminuria between acetazolamide versus placebo as measured by urinalysis.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No